CLINICAL TRIAL: NCT04156282
Title: Knot Burial Technique for Rectus Sheath Closure in Relation to Post Operative Pain in Elective Cesarean Section
Brief Title: Knot Burial Technique for Rectus Sheath Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aliaa Ibrahim Gaber Elsayed, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FWA 0000175858
Record Dates: First submitted 2019-10-14; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Intervention Model Description: we will analyze 400 candidate for elective cesarean sections, divided into two groups ,each of 200 patients according to the rectus sheath closure:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical closure. (Active Comparator): In this group, the rectus sheath closure will be done by simple running continuous sutures with the knots beneath the subcutaneous layer.
  Interventions: Procedure: classical closure
- knot burial technique (Active Comparator): The surgeon holds the left angle of the rectus sheath incision with an Allis. Using (Polyglactin 910) suture,The needle is taken from the inside outward on the upper edge.The needle is then taken lateral to the Allis and brought back into the wound by taking it through the inferior edge from outside to inside . A square knot is tied with three or four throws. The needle is then taken out of the wound through the upper edge and continuous running stitches . As the right angle is approached, the angle is held with an Allis. the suture, will be taken through the lower edge, is brought outside the wound and passed between the blades of a closed Allis before taking it inside out on the upper edge. One more bite is taken but this time just lateral to the Allis holding the angle, and the needle is brought back into the wound and to the outside between the edges of the rectus sheath. Using the loop of polyglactin held with the Allis , an Aberdeen knot is tied after removing the Allis.
  Interventions: Procedure: knot burial technique

INTERVENTIONS:
Procedure: knot burial technique — surgical suturing intervention
  Arms: knot burial technique
Procedure: classical closure — surgical suturing intervention
  Arms: classical closure.

SUMMARY:
Caesarean section is one of the most commonly performed abdominal operations on women in most countries of the world. Its rate has increased markedly in recent years, and is about 20-25% of all child-births in most developed countries.

The present study was a step to reduce postoperative pain in cesarean sections. Because of the large number of women that undergo caesarean section, even small differences in post-operative morbidity rates due to different techniques could translate into improved health and significant savings of cost and health services resources.

Closing the rectus sheath in cesarean sections with the knots pricking through the skin causes significant postoperative pain, discomfort and delayed ambulation. No comments in literature regarding the best way for closing the rectus sheath in cesarean sections.

AIM/ OBJECTIVES The aim of this study is to assess the efficacy of burying knots beneath the rectus sheath during cesarean section in reducing post operative pain and discomfort.

Study hypothesis:

In women undergoing cesarean sections may or may not burying knots beneath the rectus sheath reduce the post operative pain and discomfort.

DETAILED DESCRIPTION:
Non absorbable and delayed absorbable monofilament materials require meticulous care to prevent knot slippage.

One common problem that arises from use of these materials is the discomfort caused by the knot pricking through the skin. Although this is a common problem after cesarean section, it is often overlooked and only very few preventive techniques have been described.

This study is to assess the efficacy of burying knots beneath the rectus sheath during cesarean sections in reducing post operative pain and discomfort.

Type of Study : A randomized controlled clinical trial. Study Setting :this study will be conducted at the department of Obstetrics and Gynecology at Ain-Shams University Maternity hospital.

Study time: 2019. Study Population : The study population comprises pregnant women, fulfilling the inclusion criteria, attending to Ain Shams University Maternity Hospital, during the study period, who are planned for cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy ( more than 37 weeks of gestation ) candidate for transverse incision elective cesarean delivery

Exclusion Criteria:

* patient with BMI >30 and fat thickness >3 cm.
* patient with haemoglobin less than 10g/dL
* patient with previous history of septic wound.
* Emergency lower segment cesarean section.
* Patients complaining of premature rupture of membrane.
* Patients need intra abdominal drains post cesarean sections
* Patients with established or gestational diabetes, coagulation defects, hemodynamic instability, septicemia or chorioamnionitis.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 358 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
changing the post operative pain and discomfort | the first twenty-four hours after delivery.
  by Visual Analogue pain Scale (0) means no pain ,( 10) means sever pain.
changing the post operative pain and discomfort | one week after delivery
  by Visual Analogue pain Scale (0) means no pain ,( 10) means sever pain.
changing the post operative pain and discomfort | two weeks after delivery.
  by Visual Analogue pain Scale from ,(0) which means no pain to ( 10) means sever pain.

SECONDARY OUTCOMES:
wound assessment for suture granuloma formation | one week post operative
  by scar tissue palpation for ( presence ) or (absence) of a forming mass.
early ambulation after cesarean section | two hours after delivery
  by observation and history taking , early ambulation within two hours post operative (yes) or (no)
early breast feeding after cesarean section | two hours after delivery
  by observation and history taking, early breast feeding within two hours post operative (yes) or (no)

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa elsaid, prof.Dr, Study Director — AinShams University; Reda Mokhtar, Lecture, Study Director — AinShams University
Locations (1):
- Ahmed Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No